CLINICAL TRIAL: NCT02673385
Title: Study of the Impact of Administering t the Scale of Brazelton on the Mother's Confidence in Her Newborn Born Premature at the Approach of Returning Home
Acronym: BRAZMAMAN
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I12022
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2021-09

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Brazelton scale: Procurement across Brazelton scale
  Interventions: Other: Brazelton scale
- No test: usual care

INTERVENTIONS:
Other: Brazelton scale
  Groups: Brazelton scale

SUMMARY:
In France, the last national perinatal survey show that 6.6% of live births are premature. For these infants, transfer in Neonatology sector may result in mother-child separation can last several weeks or months. This hospital can complicate the implementation of the attachment process that allows parents to recognize their children as their own, to gain confidence in their abilities to deal with them and establish a relationship with him.

A study of mothers of premature shows the interest of the Brazelton scale to help them identify the skills their child and adjust their own behavior.

ELIGIBILITY:
Inclusion Criteria:

* Mother: over the age of 18, affiliated to a health social security.
* Newborn: born to a term of less than 36 S.A., hospitalized in neonatology, said leaving in three days.

Exclusion Criteria:

Mother :

* Legally protected
* Inability to understanding and monitoring of the protocol's terms (not master the French language, intellectual impairment, psychotic disorder ...)
* Who have had a premature child born.

New born :

* Opposition of one of the holders of parental authority to the award of the Brazelton Scale
* Having withdrawal syndromes or malformation syndromes requiring oxygen therapy, gastrostomy or nasogastric tube
* Twins and more.

Ages: 0 Weeks to 36 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Mother-child dyads whose infants were born before 36 S.A.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Score GC (Global Confidence) of the MAPS scale (Mother Assessment Baby Scale) | 2 hours

SECONDARY OUTCOMES:
Scale "EVA Anxiety" | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges Hospital, Limoges, France